CLINICAL TRIAL: NCT02206100
Title: Phase I/II Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effects of Single, Hourly-Repeating, Escalating Doses of PER977 Following a Single Subcutaneous Dose of Enoxaparin
Brief Title: PK and PD of Single, Escalating Doses of PER977 Following Enoxaparin
Acronym: PER977
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Perosphere Pharmaceuticals Inc, a wholly owned subsidiary of AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: PER977-01-003
Record Dates: First submitted 2014-06-02; First posted 2014-08-01 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: PER977; enoxaparin; anticoagulation reversal; whole blood clotting time
MeSH Terms: interventions — PER977; Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 100 mg PER977 (10 subjects); the dose may be repeated two (2) times after an approximate one (1) hour interval for a maximum total of three (3) doses
  Interventions: Drug: PER977; Drug: Placebo; Drug: enoxaparin
- Cohort 2 (Experimental): 200 mg PER977 (10 subjects); the dose may be repeated once at approximately one hour for a maximum total of two (2) doses
  Interventions: Drug: PER977; Drug: Placebo; Drug: enoxaparin
- Cohort 3 (Experimental): 300 mg PER977 (10 subjects); the dose may be repeated once at approximately one hour after the initial dose for a maximum of total of two (2) doses
  Interventions: Drug: PER977; Drug: Placebo; Drug: enoxaparin
- Cohort 4 (Experimental): 4 x 25 mg PER977 (10 subjects); study drug will be administered every 30 minutes for a total of 4 doses (cumulative dose of 100 mg PER977)
  Interventions: Drug: PER977; Drug: Placebo; Drug: enoxaparin

INTERVENTIONS:
Drug: PER977 — reversal of edoxaban-induced anticoagulation
Drug: Placebo — Reversal of edoxaban-induced anticoagulation
Drug: enoxaparin

SUMMARY:
PER977 administration following a single dose of enoxaparin

DETAILED DESCRIPTION:
Single escalating doses of PER977 from 100 to 300 mg, of 25 mg PER977 x 4 doses will be administered following administration of enoxaparin. Serial pharmacokinetic and pharmacodynamic assessments ( whole blood clotting time) will be performed. Adverse events will be monitored.

ELIGIBILITY:
Inclusion Criteria

1. Adults age 18 to 65 years, inclusive
2. Laboratory values have no clinically significant abnormalities
3. No clinically significant findings on 12-lead electrocardiogram
4. Body mass index (BMI) 18 to ≤ 27 kg/m2, inclusive
5. Male subjects agree to use appropriate contraception
6. Female subjects may be surgically sterile or post-menopausal or, if of child-bearing potential, must have a negative serum pregnancy test prior to enrollment, and must agree to use two forms of acceptable contraception for the duration of the study and for a minimum of one complete menstrual cycles or 28 days following discharge from the study.
7. Subjects must understand and agree to comply with the requirements of the study and they must be willing to sign the informed consent form indicating voluntary consent to participate in the study prior to initiation of screening or study related activities.

Exclusion Criteria:

1. History or current evidence of clinically significant disease. Current evidence of liver function tests or renal function tests greater than the upper limit of normal. The presence of Gilbert's Syndrome is acceptable. Current evidence of QTcF > normal (450±10 msec for males or 470±10 msec for females).
2. History of unexplained syncope
3. Hypersensitivity to enoxaparin sodium, thrombocytopenia with a positive in vitro test to anti-platelet antibody in the presence of enoxaparin sodium, hypersensitivity to heparin or porcine products or any other contraindication to enoxaparin
4. History of major bleeding, trauma, surgical procedure of any type, or vaginal delivery within six months prior to screening
5. History of peptic ulcer, gastrointestinal bleeding or bleeding from hemorrhoids within six months prior to screening
6. History of minor bleeding episodes such as epistaxis, or gingival bleeding within 1 month prior to screening
7. Personal or family history of clotting disorder or abnormality, excessive bleeding, thrombovascular disease or any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, or personal history of heparin-induced thrombocytopenia
8. Females with a history of dysfunctional uterine bleeding who have not undergone hysterectomy, including history of menorrhagia, metrorrhagia or polymenorrhea
9. Pregnant or breast-feeding
10. Males with a history of hormone therapy within 3 months prior to screening
11. Administration of any blood product or anticoagulant within 3 months prior to study entry or any non-steroidal anti-inflammatory drug or cyclooxygenase inhibitor within 2 weeks prior to dosing.
12. Taking any type of medication for more than 14 consecutive days within the 4 weeks prior to study entry
13. Positive serologic test for HIV, hepatitis C antibody, or hepatitis B surface antigen
14. Donation of blood or blood products within 56 days prior to screening
15. History of randomization in any prior study of PER977
16. Randomization in any study with an investigational compound or device within 30 days prior to signing informed consent
17. Active drug or alcohol dependence within the prior 12 months or any condition that, in the opinion of the Investigator, would interfere with adherence to study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 1 day
  Assessment of the number of subjects who experience adverse events and the number and type of adverse events

SECONDARY OUTCOMES:
Reversal of enoxaparin anticoagulation | 1 day
  Measurement of the degree of change in whole blood clotting time and the proportion of subjects who achieve complete or partial reversal of anticoagulation
Pharmacokinetics of enoxaparin | 1 day
  Measurement of the pharmacokinetic characteristics of enoxaparin
Pharmacokinetics of PER977 and its metabolite | 2 days
  Measurement of the pharmacokinetic characteristics of PER977 and its metabolite

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, Overland Park, Kansas, United States